CLINICAL TRIAL: NCT06119425
Title: Blood-Based Colorectal Cancer (CRC) Screening Implementation Into Clinical Practice in the Outpatient Clinical Settings in the Appalachian Highlands
Brief Title: Blood-Based Colorectal Cancer (CRC) Screening Implementation Into Clinical Practice Highlands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ballad Health (Other)
Collaborators: Guardant Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2082244-1
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2024-12

CONDITIONS: Cancer Colon
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Screening Discussion and Election (No Intervention): Patients judged to be at average risk of CRC will be engaged in a conversation about CRC risk factors and standard of care (SOC) screening options. Patients who express a desire to be screened using the SOC options will be considered part of the control group.
- Screening Selection (Experimental): Patients judged to be at average risk of CRC will be engaged in a conversation about CRC risk factors and standard of care (SOC) screening options as well as the option to be screened with a blood-based test which is not currently standard of care. Patients who express a desire to be screened using the SOC options or the blood-based non-SOC option will be considered part of the experimental group.
  Interventions: Diagnostic Test: blood-based CRC screening

INTERVENTIONS:
Diagnostic Test: blood-based CRC screening — For this study, a commercially available blood-based CRC screening test will be used. The selected test is Shield (Guardant Health, Redwood City, California, USA). The Shield test was developed, and its performance characteristics determined, by the Guardant Health Clinical Laboratory in Redwood City, California, USA, which is certified under the Clinical Laboratory Improvement Act of 1988 (CLIA) as qualified to perform high complexity clinical testing. The Shield test is currently commercially available as an laboratory developed test (LDT). Additionally, Guardant submitted the pre-market approval (PMA) application for the Shield test to the Food and Drug Administration (FDA) in March of 2023. Premarket approval (PMA) is the FDA process of scientific and regulatory review to evaluate the safety and effectiveness of medical devices. To this end, the Shield test is currently under review by the FDA.
  Arms: Screening Selection

SUMMARY:
This is a prospective implementation study that will include patients that are identified as being average risk for colorectal cancer (CRC) according to USPSTF guidelines and who have opted to be screened for CRC. The purpose of this study is to understand implementation of a noninvasive screening test in primary care and internal medicine clinical settings, and the impact on patient acceptability and adherence of CRC screening.

DETAILED DESCRIPTION:
Study Rationale This is a prospective implementation study that will include patients that are identified as being average risk for colorectal cancer (CRC) according to USPSTF guidelines and who have opted to be screened for CRC. The purpose of this study is to understand implementation of a noninvasive screening test in primary care and internal medicine clinical settings, and the impact on patient acceptability and adherence of CRC screening.

Although multiple screening options for CRC are available, participation and adherence to CRC screening remains below the national goal. CRC screening rate at the Ballad Health Mountain Laurel Internal Medicine clinic (site 1) is approximately 66%.

A blood-based test (BBT) can provide a clinically important complement to standard-of-care (SOC) screening tests and address unmet medical needs for patients, especially for those who are non-adherent with current screening modalities. There are economic and societal benefits in early detection and prevention of CRC in a broader population than the one currently up to date with screening. The unmet need for maximum participation in CRC screening could be addressed with blood-based testing.

Measuring subsequent provider experience and implementation behavior patterns involving blood based non-invasive cancer screening choices will also help to identify clinical utility of such test and implementation into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 45-84 years of age (inclusive)
* Considered by health-care providers to be "average risk" for CRC as determined by USPSTF guidelines
* If a patient opts for blood-based test, they are able and willing to provide blood samples per protocol
* Ability to understand and the willingness to participate in the study

Exclusion Criteria:

* Patients with a personal history of CRC
* Patients with a known high-risk family history of CRC precluding the patient from being average risk
* Patients with known diagnosis of inflammatory bowel disease or history of polyps
* Patients who are currently symptomatic for CRC such as: blood in the stool
* Patients with any known medical condition which, in the opinion of the investigator, should preclude enrollment into the study
* Have a recorded up to date CRC screening
* Patients with a previous abnormal colonoscopy finding who are due for surveillance.

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Opted to be screened for CRC by either SOC or study diagnostic test | 3 months
  Number of participants who agree to be screened CRC. % of participants who agree to be screened for CRC.

SECONDARY OUTCOMES:
Opted to be screened by the study diagnostic test | 3 months
  Number of participants who opted to be screened by the study diagnostic test instead of

CONTACTS AND LOCATIONS:
Overall Officials: Karen J. Elmore, MD, Principal Investigator — Ballad Health
Locations (1):
- Johnson City Medical Center, Johnson City, Tennessee, United States